CLINICAL TRIAL: NCT00175851
Title: An Open-label, Multicenter, Follow-up Trial to Evaluate the Long-term Safety and Efficacy of Seletracetam Used as Adjunctive Treatment Using a Flexible Dosing Scheme of 4 to 80 mg b.i.d. in Subjects Aged 16 Years or Older Suffering From Epilepsy
Brief Title: Open Label Trial to Study the Long-term Safety and Efficacy of Seletracetam for the Treatment of Epilepsy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Study Director, UCB
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: N01197; Not yet available
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Epilepsy
Keywords: Partial onset, primary generalized seizures, seletracetam
MeSH Terms: conditions — Epilepsy | interventions — Seletracetam

INTERVENTIONS:
Drug: Seletracetam (ucb 44212)

SUMMARY:
This is a safety and efficacy study of add-on therapy with seletracetam in epilepsy patients who have participated in a previous seletracetam study

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated IRB/IEC approved written informed consent form
* Male/female age 18 years (16 years where permitted) to 65 years
* Minimum body weight of 40 kg
* Patients having participated in a previous seletracetam study
* Female patients without childbearing potential or using a medically accepted non-hormonal contraceptive method are eligible.

Exclusion Criteria:

* Ongoing psychiatric disease other than mild controlled disorders
* Subject with clinically significant abnormalities in laboratory tests or ECG
* Poor compliance with visit schedule or medication intake in a previous seletracetam study
* Subject taking part in another clinical/pharmacological study, with the exception of seletracetam studies, in the 30 days preceding enrollment

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05

PRIMARY OUTCOMES:
Safety profile of seletracetam

SECONDARY OUTCOMES:
Reduction in seizure frequency

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Bennett, PhD, Study Director — UCB Pharma